CLINICAL TRIAL: NCT06456749
Title: An Observational, Prospective Study on the Integrated Disease Management Effectiveness of COPD and Related Comorbidities in Xishui
Brief Title: Xishui Project for IDM of COPD and Comorbidities
Status: Not yet recruiting | Type: Observational
Sponsor: China-Japan Friendship Hospital (Other)
Collaborators: Peking Union Medical College (Other); Heidelberg University (Other)
Responsible Party: Principal Investigator, Ting YANG, Professor, Associate Director of Respiratory Center, China-Japan Friendship Hospital
Other Study IDs: 2024-HX-22
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Comorbidities and Coexisting Conditions
Keywords: Effectiveness of Integrated Disease Management; Multimorbidity Management; Prosepective Cohort Study
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD patients with comorbidities: Adult patients diagnosed of stable COPD with/without diabetes and/or hypertension.4000 stable COPD patients, and among them approximately 2000 subjects with hypertension and/or type 2 diabetes complications.
  Interventions: Combination Product: Integrated Disease Management

INTERVENTIONS:
Combination Product: Integrated Disease Management — For COPD, they are encouraged to seek further cares and manage COPD on a regular basis. For smokers, they will be given a digital health intervention based on CBT. For participants with symptoms of depression or anxiety, another digital health intervention is provided. For abnormal BMI participants, a knowledge brochure will be provided and a medical worker from the township hospital will tell the harm of abnormal BMI. For hypertension and type 2 diabetes, we will actively include them into the National Essential Public Health program.

SUMMARY:
Study Population: 4000 stable COPD patients, and among them approximately 2000 subjects with hypertension and/or type 2 diabetes complications.

Design: Cohort Study Primary Objectives: The primary objective of this study is to access the effectiveness of IDM on changes in FEV1 from baseline to the 24th week visit in patients with COPD.

Statistical Analysis: We plan to compare demographic differences between groups based on whether the data conformed to normal distribution and satisfied variance chi-square, and proposed to calculate p-values using the t-test or non-parametric test for continuous data and Person's χ² or non-parametric test for categorical data. A two-sided p-value < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥40 years;
* Stable COPD patients with post-bronchodilator FEV1/FVC <70% or previously diagnosed of COPD by physicians and confirmed by PFT;
* With/without diabetes and/or hypertension;
* Permanent resident of Xishui (not expected to leave the area within 1 year).

Exclusion Criteria:

* Suffering from severe cognitive disorders or total loss of ability of daily living.
* Death.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed of stable COPD with/without diabetes and/or hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-06-17 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
FEV1 values | baseline, 24 weeks
  FEV1 values at baseline, and at week 24 in patients with COPD and in patients with COPD without diabetes or hypertension, COPD with hypertension, COPD with diabetes, and COPD with hypertension and diabetes, respectively;
Change from baseline in FEV1 values at week 24 | 24 weeks
  Change from baseline in FEV1 values at week 24 in patients with COPD and in patients with COPD without diabetes or hypertension, COPD with hypertension, COPD with diabetes, and COPD with hypertension and diabetes, respectively;

SECONDARY OUTCOMES:
Actual implementation of IDM | 48 weeks
  Actual implementation of IDM (e.g. clinical visit frequency, treatment adherence, etc.,) of over all patients, and stratified by type of comorbidities.
COPD disease outcomes | 48 weeks
  COPD disease outcomes (Life expectancy/Quality of Life/exacerbation/ mortality etc.) within week 48 and stratified by type of comorbidities.
Outpatient | 48 weeks
  Definition: Clinic or emergency utilization during the study period Functional form: Count Measurement: Medical records
Hospitalization | 48 weeks
  Definition: Hospitalization during the study period (by hospital types) Functional form: Count Measurement: Medical records
Medical expenditure | 48 weeks
  Definition: Expenditure related to healthcare Functional form: Continuous Measurement: Medical records + additional indirect expenditures recalled from questions
Quality of life (by EQ-5D-5L) | 48 weeks
  Definition: General self-rated health status Functional form: Continuous Measurement: EQ-5D instrument
Blood pressure | 48 weeks
  Definition: Systolic and diastolic blood pressure (mmHg) Functional form: Continuous Measurement: Omron portable automated sphygmomanometers
Waist circumference | 48 weeks
  Definition: Waist circumference (cm) Functional form: Continuous Measurement: Soft tape measure
Blood Glucose | 48 weeks
  Definition: glucose level in plasma Functional form: Continuous Measurement: Blood glucose meters
Body mass index | 48 weeks
  Definition: Body mass divided by the square of the body height (kg/m2) Functional form: Continuous Measurement: Calculation
Smoking Status | 48 weeks
  Definition: Do you currently smoke? Functional form: Binary/Continuous Measurement: Recall question answered by individual
Smoking Amount | 48 weeks
  Definition: If so, how many cigarettes do you smoke per day Functional form: Count Measurement: Recall question answered by individual
Alcohol | 48 weeks
  Definition: Frequency of alcohol consumption in the past 3 months Functional form: Categorical Measurement: Recall question answered by individual
Sugared consumption | 48 weeks
  Definition: Habit of sugared drink consumption Functional form: Categorical Measurement: Recall question answered by individual
Fresh Vegetable Consumption | 48 weeks
  Definition: Habit of fresh vegetables consumption Functional form: Categorical Measurement: Recall question answered by individual
Salted Vegetable Consumption | 48 weeks
  Definition: Habit of salted vegetable consumption Functional form: Categorical Measurement: Recall question answered by individual
Physical exercise | 48 weeks
  Definition: Types of physical exercise in a typical week Functional form: Categorical Measurement: Recall question answered by individual
Productivity Loss | 48 weeks
  Definition: the effect of your health problems on your ability to work and perform regular activities Functional form: Continuous Measurement: Work Productivity and Activity Impairment Questionnaire: General Health V2.0 (WPAI:GH)
Household consumption expenditures | 48 weeks
  Definition: Total household annual expenditure Functional form: Continuous Measurement: A comprehensive spectrum of expenditure categories answered by household proxy respondent
Working status | 48 weeks
  Definition: Main occupation and type Functional form: Categorical Measurement: Recall question answered by individual
Saint George Respiratory Questionnaire Score | 48 weeks
  The overall evaluation of SGRQ score

CONTACTS AND LOCATIONS:
Overall Officials: Ting Yang, MD, Principal Investigator — China-Japan Friendship Hospital; Chen Wang, MD, Study Chair — Chinese Academy of Medical Sciences and Peking Union Medical College; Simiao Chen, PhD, Principal Investigator — Chinese Academy of Medical Sciences and Peking Union Medical College